CLINICAL TRIAL: NCT00637494
Title: A Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Mifepristone vs. Placebo in the Treatment of Psychotic Symptoms in Patients With Major Depressive Disorder With Psychotic Features
Brief Title: A Study of Mifepristone vs. Placebo in the Treatment of Patients With Major Depression With Psychotic Features
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DRC recommended stopping study as it had missed its primary endpoint
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-1073-14
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Psychotic Depression; Severe Major Depression With Psychotic Features; Psychosis
Keywords: psychotic depression; major depression with psychotic features; psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Mifepristone followed by an antidepressant
  Interventions: Drug: mifepristone
- 2 (Placebo Comparator): Placebo followed by an antidepressant
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: mifepristone — 1200 mg (administered as four 300 mg tablets) once a day by mouth for the initial 7 days
  Other Names: Korlym
  Arms: 1
Drug: placebo — Tablets of identical appearance to active drug, once a day by mouth for the initial 7 days
  Other Names: control
  Arms: 2

SUMMARY:
Approximately 450 patients will be randomized to receive mifepristone or placebo for 7 days followed by antidepressant. The purpose is to compare the efficacy of mifepristone followed by antidepressant versus placebo followed by antidepressant in reducing psychotic symptoms in patients with a diagnosis of psychotic depression.

DETAILED DESCRIPTION:
Up to 450 patients with psychotic depression will be randomly assigned to receive either mifepristone or matching placebo. Patients will be assessed by the investigator or site staff during screening and on study days. A single antidepressant selected from a list of approved drugs will be administered after the administration of investigational drug. Adverse events, laboratory assessments, electrocardiograms, and physical examinations will be used to assess safety.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written consent to participate in the study prior to any study procedures and understand that they are free to withdraw from the study at any time. Patients must be able to read and understand the consent form, complete study-related procedures, and communicate with the study staff
* Have a DSM-IV TR diagnosis of Major Depressive Disorder with Psychotic Features (DSM-IV 296.24 or 296.34), and are clinically symptomatic with their illness
* Have pre-specified minimum scores on standardized psychiatric rating scales at baseline
* Have not been taking excluded medication for at least 7 days prior to randomization
* Have a negative pregnancy test
* If not postmenopausal for ≥ 2 years or surgically sterile (6 months post-surgery), must consent (patient or partner) to utilize two medically acceptable methods of contraception, one of which is a barrier method, throughout the entire study period and for 3 months after the study is completed

Exclusion Criteria:

* Have any primary psychiatric diagnosis other than psychotic depression.
* Have a major medical problem, which in the opinion of the investigator would place the patient at undue risk.
* Have undergone electroconvulsive therapy within 3 months prior to randomization
* Have had a hospitalization due to a suicide attempt within 45 days prior to randomization
* Are female and of childbearing age, and are unable or unwilling to use two medically acceptable methods of contraception during the study and for three months after study completion, one of which must be a barrier method
* Are female and are pregnant or lactating
* Are currently taking excluded medications
* Have used drugs of abuse within 30 days prior to screen, as per patient report and urine drug screen
* Have a history of active drug or alcohol abuse within 3 months or dependence within 6 months prior to screening
* Are in the opinion of the investigator at immediate risk of suicide, or at risk of harming others
* Have received investigational therapy (drug, vaccine, biological agent or device) within 6 months prior to randomization
* Have previously participated in a clinical trial of mifepristone
* Have a history of an allergic reaction to mifepristone
* Are in the investigator's opinion not appropriate for participation in the study or may not be capable of following the study schedule for any reason
* Are patients who are employees of the study unit or their family members, students who are working in the study unit, or family members of the investigator or Corcept Therapeutics

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2008-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thaddeus Block, MD, Study Director — Corcept Therapeutics
Locations (42):
- United States (42):
  - K&S Professional Research Services, LLC, Little Rock, Arkansas
  - Woodland International Research Group, Inc., Little Rock, Arkansas
  - South Coast Clinical Trials, Inc, Anaheim, California
  - Diligent Clinical Trials, Downey, California
  - Synergy Clinical Research Center, Escondido, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Pacific Research Partners, Oakland, California
  - North County Clinical Research, Oceanside, California
  - Breakthrough Clinical Trials, San Bernardino, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Cnri, Llc, San Diego, California
  - Professional Clinical Research, Inc., Aventura, Florida
  - University of Florida, Gainesville, Florida
  - Segal Institute for Clinical Research, Hollywood, Florida
  - Accurate Clinical Trials, Kissimmee, Florida
  - AMB Research Center, Miami, Florida
  - Lakeside Behavioral Health, Orlando, Florida
  - University of South Florida Dept of Psychiatry and Neurosciences, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Precise Research Centers, Flowood, Mississippi
  - Millennium Psychiatric Associate, Creve Coeur, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - CRI Lifetree, Marlton, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - Inquest Clinical Group/ Global Research Associates, Hope Mills, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Belmont Center for Comprehensive Treatment, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - FutureSearch Clinical Trials, L.P., Austin, Texas
  - Pillar Clinical Research, LLC, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Claghorn-Lesem Research Clinic, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Fein-Jennings Clinic, Inc., Houston, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeBattista C, Belanoff J, Glass S, Khan A, Horne RL, Blasey C, Carpenter LL, Alva G. Mifepristone versus placebo in the treatment of psychosis in patients with psychotic major depression. Biol Psychiatry. 2006 Dec 15;60(12):1343-9. doi: 10.1016/j.biopsych.2006.05.034. Epub 2006 Aug 4. PMID 16889757
- [Background] Flores BH, Kenna H, Keller J, Solvason HB, Schatzberg AF. Clinical and biological effects of mifepristone treatment for psychotic depression. Neuropsychopharmacology. 2006 Mar;31(3):628-36. doi: 10.1038/sj.npp.1300884. PMID 16160710
- [Background] Belanoff JK, Rothschild AJ, Cassidy F, DeBattista C, Baulieu EE, Schold C, Schatzberg AF. An open label trial of C-1073 (mifepristone) for psychotic major depression. Biol Psychiatry. 2002 Sep 1;52(5):386-92. doi: 10.1016/s0006-3223(02)01432-4. PMID 12242054
- [Background] Belanoff JK, Flores BH, Kalezhan M, Sund B, Schatzberg AF. Rapid reversal of psychotic depression using mifepristone. J Clin Psychopharmacol. 2001 Oct;21(5):516-21. doi: 10.1097/00004714-200110000-00009. PMID 11593077
- [Derived] Block TS, Kushner H, Kalin N, Nelson C, Belanoff J, Schatzberg A. Combined Analysis of Mifepristone for Psychotic Depression: Plasma Levels Associated With Clinical Response. Biol Psychiatry. 2018 Jul 1;84(1):46-54. doi: 10.1016/j.biopsych.2018.01.008. Epub 2018 Jan 31. PMID 29523415
- See also: Corcept Therapeutics — http://www.corcept.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Mifepristone 1200 mg/Day: Mifepristone 1200 mg/day on Days 1-7 and a single-study approved antidepressant on Days 8-56
- Matching Placebo: Matching placebo on Days 1-7 and a single-study approved antidepressant on Days 8-56
Period: Overall Study
Arm/Group | Mifepristone 1200 mg/Day | Matching Placebo
Started | 141 | 151
Completed | 109 | 108
Not Completed | 32 | 43

BASELINE CHARACTERISTICS:
Groups:
- Mifepristone Followed by an Antidepressant: Mifepristone 1200 mg/day on Days 1-7 and a single-study approved antidepressant on Days 8-56
- Total: Total of all reporting groups
Arm/Group | Mifepristone Followed by an Antidepressant | Matching Placebo | Total
Number analyzed (Participants) | 141 | 151 | 292
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 141 | 147 | 288
  >=65 years | 0 | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (9.0) | 47.0 (9.5) | 46.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 85 | 161
  Male | 65 | 66 | 131
Region of Enrollment [Number; unit: participants]
  United States | 141 | 151 | 292

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Mifepristone vs. Placebo Treated Patients With at Least a 50% Reduction From Baseline in Brief Psychiatric Rating Scale-Positive Symptom Subscale (BPRS-PSS) at Days 7 and 56
Description: Response as measured by 50% reduction in psychosis at Days 7 and 56 was compared between the group administered placebo and the group administered mifepristone
Time Frame: 56 days
Measure: Number; unit: participants
Groups:
- Active: Mifepristone followed by an antidepressant
  mifepristone: 1200 mg (administered as four 300 mg tablets) once a day by mouth for the initial 7 days
- Placebo: Placebo followed by an antidepressant
  placebo: Tablets of identical appearance to active drug, once a day by mouth for the initial 7 days
Arm/Group | Active | Placebo
Number analyzed (Participants) | 141 | 151
participants | 51 | 48

2. Secondary Outcome: Proportion of Mifepristone Treated Patients With Plasma Drug Concentrations Equal to or Above 1637 ng/mL vs. Placebo Treated Patients Who Achieve a ≤ 50% Reduction in BPRS-PSS at Days 7 and 56
Description: Response as measured by 50% reduction in psychosis at Days 7 and 56 was compared between the group administered placebo and the group who achieved a sufficiently high plasma level of mifepristone
Time Frame: 56 days
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 94 | 151
participants | 37 | 48

ADVERSE EVENTS:
Arm/Group | Mifepristone 1200 mg/Day | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 3/141 | 4/151
Other Adverse Events (participants affected / at risk) | 115/141 | 103/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone 1200 mg/Day (N=141) | Matching Placebo (N=151)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Psychotic Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Nervous system disorders) | 1 (1) | 2 (2)
Suicidal Ideation (Nervous system disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone 1200 mg/Day (N=141) | Matching Placebo (N=151)
Nausea (Gastrointestinal disorders) | 25 (35) | 19 (20)
Constipation (Gastrointestinal disorders) | 17 (20) | 14 (16)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 14 (15)
Dry Mouth (Gastrointestinal disorders) | 15 (15) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 14 (16) | 9 (10)
Vomiting (Gastrointestinal disorders) | 11 (11) | 8 (8)
Abdominal Pain (Gastrointestinal disorders) | 7 (7) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9) | 3 (3)
Headache (Nervous system disorders) | 33 (41) | 29 (32)
Dizziness (Nervous system disorders) | 11 (11) | 9 (9)
Insomnia (Psychiatric disorders) | 8 (9) | 16 (16)
Anxiety (Psychiatric disorders) | 8 (8) | 9 (11)
Fatigue (General disorders) | 9 (16) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 6 (6)
Pollakiuria (Renal and urinary disorders) | 12 (15) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other